CLINICAL TRIAL: NCT04278235
Title: Expanded Access to Elezanumab
Status: Available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C20-203; C20-284 (Other Grant/Funding Number: Abbvie); C20-285 (Other Grant/Funding Number: Abbvie)
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-04

CONDITIONS: Acute Spinal Cord Injury (SCI)
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: interventions — elezanumab

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Drug: Elezanumab — Solution for intravenous (IV) infusion
  Other Names: ABT-555

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to Elezanumab prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Exclusion Criteria:

* There are other suitable treatment options.
* The participant qualifies for ongoing clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie